CLINICAL TRIAL: NCT02171273
Title: Impact of Chronic Circadian Disruption vs. Chronic Sleep Restriction on Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Charles Andrew Czeisler, MD, PhD, Baldino Professor of Sleep Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2014-P-000243; 2P01AG009975-16A1 (NIH)
Record Dates: First submitted 2014-06-16; First posted 2014-06-24 (Estimated); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Aging; Sleep Restriction; Circadian Disruption
Keywords: Sleep; Aging; Metabolism; Circadian; Genetic; Alertness

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Chronic circadian disruption (Experimental): Following a baseline of adequate time in bed, study participants will spend 3 weeks on a daily jet-lag schedule (where each day is longer than 24 hours).
  Interventions: Behavioral: Circadian Disruption
- Chronic sleep restriction (Experimental): Following a baseline of adequate time in bed, study participants will have a shortened opportunity for sleep during each 24-hour day (for three weeks).
  Interventions: Behavioral: Sleep Restriction
- Control (sleep extension) (Active Comparator): Following a baseline of adequate time in bed, study participants will continue to have adequate time in bed and opportunity for sleep during each 24-hour day, for 3 weeks.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Circadian Disruption — Following a baseline of adequate time in bed, study participants will spend 3 weeks on a daily jet-lag schedule (where each day is longer than 24 hours).
  Arms: Chronic circadian disruption
Behavioral: Sleep Restriction — Following a baseline of adequate time in bed, study participants will have a shortened opportunity for sleep during each 24-hour day (for three weeks).
  Arms: Chronic sleep restriction
Behavioral: Control — Following a baseline of adequate time in bed, study participants will continue to have adequate time in bed and opportunity for sleep during each 24-hour day, for 3 weeks.
  Arms: Control (sleep extension)

SUMMARY:
The overall objectives of the proposed study are to examine the consequences of chronic circadian disruption and chronic sleep restriction on metabolic function in healthy adults.

DETAILED DESCRIPTION:
It has long been recognized that sleep patterns change with age. A common feature of aging is the advance of the timing of sleep to earlier hours, often earlier than desired. These age-related changes are found in even healthy individuals who are not taking medications and who are free from sleep disorders. In addition to these sleep disturbances, many older individuals curtail their sleep voluntarily, reporting similar rates of sleep restriction (sleeping less than 7 or less than 6 hours per night) when compared to young adults. Whether voluntary or not, insufficient sleep has medical, safety and metabolic consequences. In fact, converging evidence in young adults suggests that sleep restriction per se may impair metabolism, and that reduced sleep duration is associated with weight gain, obesity, diabetes, cardiovascular disease, and mortality. An understanding of how the circadian and sleep homeostatic neurobiological processes responds to increasing homeostatic sleep pressure, and the effects of sleep restriction on metabolism at different ages, should provide information on the regulation of sleep and metabolism in aging, as well as direction for future treatments. In the present study, we will study the separate impacts of chronic sleep restriction (while minimizing circadian disruption) and chronic circadian disruption (while minimizing sleep disruption) and a poor diet on metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults with conventional and regular sleep-wake timing
* Non-smokers
* Completion of medical, psychological, and sleep screening tests
* Able to spend 37 consecutive days/nights in the laboratory

Exclusion Criteria:

* History of neurological or psychiatric disorder
* History of sleep disorder or regular use of sleep-promoting medication
* Current prescription, herbal, or over-the-counter medication use
* Traveling across 2 or more time zones within past 3 months
* Donating blood within past 8 weeks
* Worked night or rotating shift work within past 3 years
* Hearing impairment
* Drug or alcohol dependency

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2014-03-31 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Change in insulin sensitivity | Baseline day 3, at 1 week and at 3 weeks of exposure, and 1 week into recovery
  Euglycemic hyperinsulinemic clamp-assessed measure of insulin sensitivity
Changes in glucose levels after standardized meal | Baseline day 2, daily throughout 1st and 3rd weeks of exposure, and 1 week into recovery
  Frequent blood samples during and after standardized meal (breakfast), response of blood glucose levels
Change in insulin levels after standardized meal | Baseline day 2, daily throughout 1st and 3rd weeks of exposure, and 1 week into recovery
  Frequent blood samples during and after standardized meal (breakfast)
Change in 24h profiles of leptin | Baseline day 2, during acute circadian misalignment (exposure day 3), and acute realignment (exposure day 7)
  Hourly blood samples for 24 hours
Change in 24h profiles of cortisol | Baseline day 2, at 3 weeks of exposure, and 1 week into recovery
  Hourly blood samples for 24 hours

SECONDARY OUTCOMES:
Change in resting metabolic rate | Baseline days 2 and 3, daily throughout 1st and 3rd weeks of exposure, and 1 week into recovery
  Indirect calorimetry, daily body weight, core body temperature
Change in circadian phase and/or period | Continuous throughout the 3-day baseline, 3-week exposure, and 1-week recovery
  Via measurement of core body temperature and melatonin (salivary and plasma)
Changes in sleep/wake architecture and brain electrical activity | Continuous throughout the 3-day baseline, 3-week exposure, and 1-week recovery
  Polysomnography during sleep and wake
Change in neurocognitive performance | Daily throughout the 3-day baseline, 3-week exposure, and 1-week recovery
  Cognitive test battery presented via computer interface
Changes in perception of pain, hunger and sleepiness | Daily throughout the 3-day baseline, 3-week exposure, and 1-week recovery
  Daily questionnaires
Change in inflammatory markers and wake-time hormone levels | Baseline days 2 and 3, daily throughout 1st and 3rd weeks of exposure, and 1 week into recovery
  Measurements on fasted blood samples
Changes in daily patterns of gene expression, epigenetic or proteomic markers | Baseline day 2, at 1 week and at 3 weeks of exposure, and 1 week into recovery
  Blood samples collected every 4 hours for 48 hours
Changes in measures of sympathovagal balance and autonomic function | Baseline day 3, at 1 week and at 3 weeks of exposure, and 1 week into recovery
  EKG, urinary catecholamines, fasting and postprandial blood samples for cortisol, epinephrine and norepinephrine
Change in nutrient absorption | Daily throughout the 3-day baseline, last 3 days of the 3-week exposure, and last three days of the 1-week recovery
  Bomb calorimetry on stool samples

CONTACTS AND LOCATIONS:
Overall Officials: Charles A Czeisler, PhD, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Xin Q, Yuan RK, Zitting KM, Wang W, Purcell SM, Vujovic N, Ronda JM, Quan SF, Williams JS, Buxton OM, Duffy JF, Czeisler CA. Impact of chronic sleep restriction on sleep continuity, sleep structure, and neurobehavioral performance. Sleep. 2022 Jul 11;45(7):zsac046. doi: 10.1093/sleep/zsac046. PMID 35218665